CLINICAL TRIAL: NCT01263639
Title: Improving Patient Satisfaction in the Orthopaedic Trauma Population
Brief Title: Improving Patient Satisfaction Improving Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Brent Joseph Morris, Orthopaedic Resident, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: Patient Satisfaction; Clinical Trial (Other Grant/Funding Number: National Center for Advancing Translational Sciences (grant 2 UL1 TR000445-06).)
Record Dates: First submitted 2010-12-16; First posted 2010-12-21 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-06

CONDITIONS: Satisfaction; Trauma
Keywords: patient satisfaction; patient-physician relationship; orthopaedic trauma
MeSH Terms: conditions — Personal Satisfaction; Wounds and Injuries; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group, biosketch card (Experimental): The investigators aim to improve the patient-physician relationship and improve patient satisfaction by providing a biosketch card of the attending orthopaedic trauma surgeon to the patient. The biosketch card will include a picture of the attending orthopaedic surgeon with a brief synopsis of his or her: education background, specialty, surgical interests, research interests, and other interests including hobbies.
  Interventions: Other: Orthopaedic Attending Biosketch Card
- Control group, standard care (Active Comparator): The "intervention" group will receive an attending photo/biosketch card within 24 hours of admission while the control group will not. The control group will receive the usual/standard care as provided to all orthopaedic trauma admission patients without receiving a biosketch card.
  Interventions: Other: Standard of care - No biosketch card

INTERVENTIONS:
Other: Orthopaedic Attending Biosketch Card — The "intervention" group will receive an attending photo/biosketch card within 24 hours of admission while the control group will not. The biosketch card will include a picture of the attending orthopaedic surgeon with a brief synopsis of his or her: education background, specialty, surgical interests, research interests, and other interests including hobbies.
  Arms: Intervention Group, biosketch card
Other: Standard of care - No biosketch card — Standard of care
  Arms: Control group, standard care

SUMMARY:
Objectives: Patient satisfaction is a key determinant of the quality of care and an important component of pay for performance metrics. The purpose of this study was to evaluate the impact of a simple intervention aimed to increase patients' understanding of their orthopaedic trauma surgeon and improve patient satisfaction with the overall quality of inpatient care delivered by the attending surgeon.

Design: Prospective quality improvement initiative using a randomized intervention.

Setting: Level 1 academic trauma center.

Patients/Participants: Two hundred twelve patients were eligible; 100 patients were randomized to the intervention group, and 112 patients were randomized to the control group. Overall, 76 patients could be reached for follow-up satisfaction survey, including 34 patients in the intervention group and 42 patients in the control group.

Intervention: Patients randomized to the intervention group received an attending biosketch card, which included a picture of the attending orthopaedic surgeon with a brief synopsis of his educational background, specialty, surgical interests, and research interests.

Main Outcome Measures: Our primary outcome measure was a patient satisfaction survey assessing patients' rating of the overall quality of inpatient care delivered by the attending surgeon.

DETAILED DESCRIPTION:
Patient satisfaction is a key determinant of the quality of care and an important component of pay for performance metrics. The Centers for Medicare & Medicaid Services (CMS) Hospital Inpatient Value-Based Purchasing Program implemented value-based incentive payments that link Medicare reimbursements to patient satisfaction and physician surveys completed by patients.1 There is a paucity of data in the orthopaedic literature assessing patient satisfaction, especially regarding patients with orthopaedic trauma. Surprisingly, up to 90% of medical inpatients are unable to correctly name their treating physician when asked to identify the physician in charge of his or her care at the time of discharge.2-4 The orthopaedic trauma patient population is even more challenging due to traumatic injuries warranting inpatient surgery in the acute setting as opposed to elective surgeries or medical admissions. Admissions from the emergency department have been associated with a decreased ability of patients to identify their treating physician. 3 Furthermore, the acuity of these injuries does not always permit patients and surgeons to establish a strong patient-physician relationship before the surgery. Patient-physician communication is integral to improving clinical relationships and improving patient satisfaction.5,6 Surgeons exhibit a tendency to focus on operative quality and outcomes, whereas patients place greater value on the surgeon-patient interaction.7,8 Establishing rapport and a strong patient-physician relationship in the acute trauma setting is challenging but being able to recognize the name and face of the attending orthopaedic surgeon is a critical step in the communication chain. The presence of attending physician photographs in patient rooms has been associated with a significant improvement in the ability to correctly identify the attending physician and is associated with improved patient satisfaction.4,9 The purpose of this prospective quality improvement study was to evaluate the impact of a simple intervention aimed to increase patient recognition of the attending orthopaedic trauma surgeon and improve patient satisfaction with the overall quality of care delivered by the attending surgeon during the inpatient stay. Patients randomized to intervention group received an attending biosketch card, whereas patients randomized to the control group did not receive a card. Our hypothesis was that the patients in the intervention group (received attending biosketch card) would have higher patient satisfaction scores regarding the overall care provided by his or her attending orthopaedic trauma surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100 year old patients
* English speaking
* Admitted to the orthopaedic trauma surgery service
* Isolated orthopaedic injury requiring orthopaedic surgery on the same admission

Exclusion Criteria:

* <18 years old
* traumatic brain injury
* Admission greater than 7 days
* patients with prior orthopaedic trauma injuries treated at Vanderbilt University Medical Center (VUMC)
* patients with prior patient patient-physician relationship with orthopaedic trauma attending
* visually impaired patients
* intubated/sedated patients
* intoxicated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent J Morris, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderiblt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Morris BJ, Richards JE, Archer KR, Lasater M, Rabalais D, Sethi MK, Jahangir AA. Improving patient satisfaction in the orthopaedic trauma population. J Orthop Trauma. 2014 Apr;28(4):e80-4. doi: 10.1097/01.bot.0000435604.75873.ba. PMID 24158181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2011 to December 2011. All patients were admitted from the ER to the orthopaedic trauma service and had operative injuries requiring surgery on the same admission.
Period: Overall Study
Arm/Group | Intervention Group, Biosketch Card | Control Group, Standard Care
Started | 107 | 121
Completed | 34 | 42
Not Completed | 73 | 79
Not completed — Lost to Follow-up | 66 | 70
Not completed — Exclusion =Admission greater than 7 days | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group, Biosketch Card | Control Group, Standard Care | Total
Number analyzed (Participants) | 107 | 121 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 80 | 88 | 168
  >=65 years | 21 | 27 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (17.3) | 41.9 (17.1) | 42.3 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 52 | 95
  Male | 64 | 69 | 133
Region of Enrollment [Number; unit: participants]
  United States | 107 | 121 | 228

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction as Measured by Giving an "Excellent" Score on a 5-point Rating
Description: Within 2 weeks of discharge from the hospital, but before the patient's first clinic visit, each group will be called by the Professional Resource Group as part of regular quality improvement by the Vanderbilt Medical Center Department of Strategic Development. The patients will be asked a series of questions aimed at determining overall patient satisfaction based on interactions with the attending orthopaedic trauma surgeon.
Time Frame: within 2 weeks of discharge and before first clinic appointment
Measure: Number; unit: participants
Arm/Group | Intervention Group, Biosketch Card | Control Group, Standard Care
Number analyzed (Participants) | 34 | 42
participants | 25 | 22

ADVERSE EVENTS:
Arm/Group | Intervention Group, Biosketch Card | Control Group, Standard Care
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/112
Other Adverse Events (participants affected / at risk) | 0/100 | 0/112

LIMITATIONS AND CAVEATS:
No adverse events. Limitations included poor patient follow-up due to poor patient participation with telephone call surveys.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No